CLINICAL TRIAL: NCT06343766
Title: Polymorphisms in ENAM, AMBN, and KLK4 Predispose Egyptian Adults to Dental Caries: A Cross-Sectional Study
Brief Title: Polymorphisms in ENAM, AMBN, and KLK4 Contribute to DCS.
Status: Completed | Type: Observational
Sponsor: Amina Fouad Farag (Other)
Responsible Party: Sponsor-Investigator, Amina Fouad Farag, Associate Professor of Oral and Maxillofacial Pathology, Oral Pathology Department, Faculty of Dentistry, October 6 University
Organization: October 6 University (Other)
Other Study IDs: RECO6U/24-2022
Record Dates: First submitted 2024-03-19; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Dental Caries Secondary to Polymorphisms; Polymorphisms in Enamel Encoding Genes
Keywords: Enamelin (ENAM); Ameloblastin (AMBN); Tuftelin 1 (TUFT1); Kallikrein-related peptidase-4 (KLK4); Dental caries; Polymorphisms
MeSH Terms: conditions — Dental Caries | interventions — Genotype; Diagnosis, Oral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA was collected from all participants using buccal swabs provided in the Sigma® Cheek Cell Collection Kit in this study. These swabs were gently rubbed on both sides of the buccal mucosa ten times. After removing the plastic sticks from the swabs, the collected swabs were placed in 1.5-ml Eppendorf tubes. These tubes were then stored at +4 °C until genomic DNA extraction. Following a brief centrifugation, DNA purification was performed following the manufacturer's instructions. The purified DNA samples were subsequently stored at -21 °C for future analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Caries-susceptible group
  Interventions: Genetic: DNA collation and genotyping
- Control group: Caries-resistant group
  Interventions: Genetic: DNA collation and genotyping

INTERVENTIONS:
Genetic: DNA collation and genotyping — DNA collation and genotyping of specific genes ENAM rs3796703, AMBN rs4694075), TUFT1 rs78802584 and KLK4 rs2242670 through PCR and sequencing for various SNPs
  Dental examinations by comparing dental covariates such as the number of DMF-T index, presence of biofilm, gingivitis, fluorosis, and detection of interproximal caries with caries progression.
  Other Names: Dental examinations

SUMMARY:
A Cross-Sectional Study aims to shed light on potential genetic determinants influencing dental caries susceptibility within this demographic and significantly understanding of genetic factors associated with dental caries, particularly within the context of the Egyptian population, providing valuable insights into the genetic aspects of oral health. The research methodology involved a comprehensive examination of these polymorphic loci ENAM, AMBN, TUFT1 and KLK4 and their prevalence, employing rigorous statistical analyses to establish potential correlations between these genetic variants and susceptibility to dental caries.

DETAILED DESCRIPTION:
The research investigates the distributional discrepancies of specific polymorphic loci ENAM rs3796703, AMBN rs4694075, TUFT1 rs13236243, and KLK4 rs2242670-within the Egyptian population as correlatives and causatives of dental caries susceptibility through the genotyping of enamelin (ENAM rs3796703), ameloblastin (AMBN rs4694075), tuftelin 1 (TUFT1 rs78802584), and kallikrein 4 (KLK4 rs2242670) in 132 adults (males = 74, females = 58) and 72 controls (males = 40, females = 32) referred from various Egyptian hospitals. For each participant, the number of decayed, missing, and filled teeth was charted, and the presence of biofilm/gingivitis/fluorosis was assessed. Bitewing radiographs were taken to detect interproximal caries. In addition, statistical analysis was conducted using Chi-square test, odds ratios, and corresponding P-values.

ELIGIBILITY:
Inclusion Criteria:

* Presence of dental caries or decay in form of discoloration, cavities, or visible enamel softening suggestive of potential caries (Caries-susceptible group)
* Caries-free patients as control group (Caries-resistant group)

Exclusion Criteria:

* The presence of white spots or fluorosis, indicating enamel defects or demineralization, required exclusion from the study.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients presented to Operative Dentistry Department, Faculty of Dentistry and Outpatient Clinics of University Hospital of October 6 University and referred from various Egyptian hospitals in Greater Cairo, Egypt
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Polymorphisms in genes associated with enamel formation and mineralization and dental caries susceptibility. | Done immediately following completion of assessment for eligibility of enrolment in the present study
  Potential role of alleles or genotypes of enamel encoding genes such as ENAM, AMBN, TUFT1 and KLK4 in the caries-susceptible group and in the caries-resistant group using PCR and sequencing for various SNPs

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M. Negm, PhD, Principal Investigator — Faculty of Dentistry, October 6 University, Giza, Egypt; +201222323200; Hassannegm.dent@o6u.edu.eg; Rania R. Omar, PhD, Principal Investigator — Faculty of Dentistry, October 6 University, Giza, Egypt; rania.rashad@dentistry.cu.edu.eg; Amina F. Farag, PhD, Principal Investigator — Faculty of Dentistry, October 6 University, Giza, Egypt; AminaFouadFarag.dent@o6u.edu.eg
Locations (1):
- Faculty of Dentistry, October 6 University, Giza, Egypt